CLINICAL TRIAL: NCT02453490
Title: The Second Affiliated Hospital of Zhejiang University
Brief Title: Compare Efficacy and Safety of Raltitrexed-based and 5fu-based Neoadjuvant Chemotherapy for Colorectal Liver Metastasis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficultly recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, the Second Affiliated Hospital of Zhejiang University, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRCLM-01
Record Dates: First submitted 2015-05-17; First posted 2015-05-25 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer; Liver Metastasis
Keywords: Colorectal Cancer; liver metastasis; neoadjuvant chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltitrexed-based chemotherapy (Experimental): Raltitrexed plus Oxaliplatin/Raltitrexed plus Irinotecan
  Interventions: Drug: Raltitrexed-based chemotherapy
- 5-fluorouracil-based chemotherapy (Active Comparator): 5-fluorouracil plus Oxaliplatin/5-fluorouracil plus Irinotecan
  Interventions: Drug: 5-fluorouracil-based chemotherapy

INTERVENTIONS:
Drug: Raltitrexed-based chemotherapy — Raltitrexed: 2.0mg,iv,15min,d1,Oxaliplatin:85mg/m2 iv,d1, q2w
  Other Names: RTXOX
  Arms: Raltitrexed-based chemotherapy
Drug: Raltitrexed-based chemotherapy — Raltitrexed: 2.0mg,iv,15min,d1,Irinotecan:180mg/m2 iv,d1, q2w
  Other Names: RTXIRI
  Arms: Raltitrexed-based chemotherapy
Drug: 5-fluorouracil-based chemotherapy — 5-fluorouracil:400mg/m2,ivp,2h,d1,1200mg/m2/d*2d(2400mg/m2,iv46-48h); Oxaliplatin:85mg/m2 iv,d1,q2w
  Other Names: mFOLFOX6
  Arms: 5-fluorouracil-based chemotherapy
Drug: 5-fluorouracil-based chemotherapy — 5-fluorouracil: 400mg/m2,ivp,2h,d1,1200mg/m2/d*2d(2400mg/m2,iv46-48h); Irinotecan:180mg/m2 d1, iv,q2w
  Other Names: FOLFIRI
  Arms: 5-fluorouracil-based chemotherapy

SUMMARY:
This study is a multicenter ,randomization, open control study to evaluate the efficacy and safety of Raltitrexed-based chemotherapy and 5-fluorouracil-based chemotherapy in the peri-operative treatment of patients with Liver Metastasis From colorectal cancer (CRC).

DETAILED DESCRIPTION:
The contrast analysis is separately done on Raltitrexed plus oxaliplatin and 5-fluorouracil plus oxaliplatin;Raltitrexed plus irinotecan and 5-fluorouracil plus irinotecan.To investigate the objective response rate,the R0 resection rate, the early tumor shrinkage （ETS）and depth of response(DPR) and the safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed chinese colorectal cancer patients and imaging detection confirmed liver metastasis
2. previously no treatment for liver metastasis or Primary tumor had been removed and last additional chemotherapy over one year
3. Age of≥18 and ≤75
4. Adequate organ functions, as determined by normal bone marrow function (absolute neutrophil count2 x 109/L, platelets 100 x 109/L, White blood cells 4 x 109/L), liver function (serum bilirubin ≤ 2.5 x ULN, serum transaminases ≤2. 5x ULN)
5. ECOG≤1
6. Life Expectancy>6months
7. Signed written informed consent
8. Expected adequacy of follow-up

Exclusion Criteria:

1. Lesion is too small to assess by imaging
2. Extrahepatic metastases
3. Any anticancer chemotherapy in development within 4 weeks prior to study entry
4. Concurrent uncontrolled illness such as infection
5. Be allergic to medicines in the study
6. Pregnant or nursing patients
7. Fertile women (< 2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception.
8. Not willing or incapable to comply with all study visits and assessments
9. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that puts the patient at high risk for treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2015-10-11 (Actual); Primary Completion 2018-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 38 months

SECONDARY OUTCOMES:
R0 resection rate of liver | 38 months

OTHER OUTCOMES:
The side effects of the treatment | 38 months
The early tumor shrinkage （ETS）and depth of response(DPR) | 38 months

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ke-Feng, PHD/MD, Study Chair — Zhejiang University
Locations (9):
- China (9):
  - The Affiliated Tumor Hospital of Zhongshan University, Guangzhou, Guangdong
  - Wuhan Union Hospital, Wuhan, Hubei
  - Zhongnan Hospital Affiliated to Wuhan University, Wuhan, Hubei
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Second Affiliated Hospitalof Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jinhua People's Hospital, Jinhua, Zhejiang
  - The second hospital of Ningbo City, Ningbo, Zhejiang